CLINICAL TRIAL: NCT04008212
Title: Feasibility of Computer-assisted Aortic and Iliac Endovascular Procedures With Mobile C-arm
Brief Title: Fusion Imaging for EVAR With Mobile C-arm
Acronym: FUTUR
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC15_3020
Record Dates: First submitted 2019-07-02; First posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Fusion Imaging for EVAR

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- EVAR aneurysm
  Interventions: Other: Fusion imaging
- Stenosis
  Interventions: Other: Fusion imaging

INTERVENTIONS:
Other: Fusion imaging — Fusion imaging during aortic endovascular procedures with a mobile C-arm through the use of the EndoNaut® angio-navigation station

SUMMARY:
Fusion imaging is a technique that facilitates endovascular navigation but is only available in hybrid rooms. The goal of this study is to evaluate the feasibility of fusion imaging with a mobile C-arm in a conventional operating room through the use of an angio-navigation station.

DETAILED DESCRIPTION:
The study include all patients who underwent an aortic stent graft procedure in a conventional operating room with a mobile flat-panel detector (Cios Alpha, Siemens) connected to an angio-navigation station (EndoNaut, Therenva). The intention is to perform preoperative 3D CT/perioperative 2D fluoroscopy fusion Imaging using an automatic registration process. Registration is considered successful when the software was able to correctly overlay preoperative 3D vascular structures onto the fluoroscopy image. For EVAR, contrast dose, operation and fluoroscopy time were compared to those of a control group drawn from the department's database who underwent a procedure with a C-arm image intensifier.

ELIGIBILITY:
Inclusion Criteria:

Patients eligible for endovascular treatment of aneurysm disease of the aorta. Procedure performed in a conventional operating room equipped with a mobile flat-panel detector (30´30 cm) (Cios-Alpha, Siemens®, Munich, Germany) and a floating table.

Patients who received written and verbal information about the protocol and did not object to participating in the trial.

Exclusion Criteria:

Patients who also required a conventional surgical revascularisation procedure or who required an endovascular revascularisation procedure in another site.

Patients who underwent MR angiography during preoperative evaluation. Non-analysable CT angiogram (no or poor injection). Procedure performed in a hybrid room or in an operating room not equipped with a mobile flat-panel detector.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients eligible for endovascular treatment of aneurysm disease of the aorta.
Sampling Method: Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-07-19 (Actual); Study Completion 2018-02-02 (Actual)

PRIMARY OUTCOMES:
Feasibility of fusion imaging | 6 months
  To evaluate the feasibility of fusion imaging during aortic endovascular procedures with a mobile C-arm through the use of the EndoNaut® angio-navigation station

IPD SHARING:
Plan to Share IPD: Undecided